CLINICAL TRIAL: NCT06654700
Title: A Randomized, Double-blind Phase III Clinical Trial to Evaluate the Lot-to-lot Consistency of Three Consecutive Batches of Recombinant Herpes Zoster Vaccine (CHO Cell) Produced At a Commercial Scale in Subjects Aged 40 Years and Older.
Brief Title: Phase III Clinical Trial of Lot-to-lot Consistency of Recombinant Herpes Zoster Vaccine (CHO Cell).
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: MAXVAX Biotechnology Limited Liability Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MKKCT-100-004
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Herpes Zoster
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Herpes Zoster vaccine（Commercial-scale batch 1 group） (Experimental): Subjects will receive Recombinant Zoster Vaccine (CHO cell) according to a 0, 2-month schedule
  Interventions: Biological: Recombinant Zoster Vaccine (CHO Cell)
- Herpes Zoster vaccine（Commercial-scale batch 2 groups） (Experimental): Subjects will receive Recombinant Zoster Vaccine (CHO cell) according to a 0, 2-month schedule
  Interventions: Biological: Recombinant Zoster Vaccine (CHO Cell)
- Herpes Zoster vaccine（Commercial-scale batch 3 groups） (Experimental): Subjects will receive Recombinant Zoster Vaccine (CHO cell) according to a 0, 2-month schedule
  Interventions: Biological: Recombinant Zoster Vaccine (CHO Cell)

INTERVENTIONS:
Biological: Recombinant Zoster Vaccine (CHO Cell) — 0.5 mL per dose, containing a total of 50 µg recombinant varicella zoster virus glycoprotein E, adjuvanted with MA105. Intramuscular injection

SUMMARY:
To evaluate the lot-to lot consistency of three batches of recombinant herpes zoster vaccine (CHO cell) produced on a commercial scale in subjects aged 40 years and older after receiving 2 doses on a 0, 2 month schedule.

DETAILED DESCRIPTION:
A total of 1200 subjects aged 40 years and older were randomly assigned in a 1:1:1 ratio to three commercial-scale batches (batch 1, batch 2, Batch 3) , with 400 subjects in each group. To demonstrate lot-to-lot consistency in terms of anti-gE antibody GMC between three production lots of the HZ vaccine one month after the second dose.

ELIGIBILITY:
Inclusion Criteria:

1. A male or female permanent resident aged 40 years and older at enrollment, with valid identity;
2. Subjects voluntarily agree to participate in the study and signed an informed consent;
3. Be able to understand clinical trials, participate in all scheduled visits and comply with the protocol requirements(e.g. completion of the diary cards/questionnaires, return for follow-up visits, have regular contact to allow evaluation during the study);
4. Women of childbearing potential plan to avoid pregnancy and are willing to use effective contraception(e.g. oral contraceptive pills, injectable progestogen, percutaneous contraceptive patches, implants of levonorgestrel, intrauterine device, female and male sterilization or abstinence) within 12 months after the last vaccination, and the uses of the rhythm method alone, withdrawal alone, and emergency contraception, are not acceptable.

Exclusion Criteria:

1. Axillary temperature > 37.0°C on the day of vaccination or acute illness;
2. Current or history of herpes zoster;
3. Previous vaccination against varicella or herpes zoster (either registered product or participation in a previous vaccine study);
4. Pregnant (urine pregnancy test was positive) or lactating female;
5. Receipt of live vaccine within 28 days, or any other vaccine within 14 days prior to vaccination;
6. Receipt of immunoglobulin or intravenous immunoglobulin during 3 months before vaccination, or planned receipt 1 month post the last vaccination;
7. Acute diseases(such as acute upper respiratory tract infection with fever, cough, sore throat) or acute exacerbation of chronic disease within 3 days before vaccination;
8. Receipt of antipyretic, analgesic and allergy drugs within 3 days before vaccination, except enteric-coated aspirin for cardiovascular diseases prevention;
9. A known allergy to any components of the study vaccine, or history of severe allergy (e.g. Anaphylactic shock, allergic laryngeal edema, anaphylactoid purpura, thrombocytopenic purpura, Arthus reaction, severe urticaria) to any previous vaccination;
10. Allergy to aminoglycoside antibiotics;
11. History of convulsions, epilepsy, congenital brain dysplasia, mental illness or family history, or history of brain nerve tissue damage due to other severe neurological disorders(e.g. brain tumor, cerebral hemorrhage, cerebral infarction, brain infection disease, chemical drug poisoning);
12. Asplenia or functional asplenia, or splenectomy caused by any condition;
13. Primary or secondary impairment of immune function, diagnosed congenital or acquired immunodeficiency, human immunodeficiency virus (HIV) infection, lymphoma, leukemia, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease or other autoimmune diseases;
14. Receipt of Immunosuppressive therapy(such as long-term use of systemic glucocorticoid ≥14 days, ≥20mg/day prednisone or equivalent dose) or long-acting immune-modifying drugs(e.g. Infliximab) during the period starting 6 months before vaccination or planned administration 1 month after the last vaccination, but topical steroids(e.g. ointment, eye drops, inhalants, nasal sprays) that do not exceed the dosage recommended in the instructions or have any systemic signs are acceptable;
15. Patients with severe chronic diseases, including but not limited to severe cardiovascular diseases (pulmonary heart disease, pulmonary edema), severe liver and kidney diseases, and diabetes mellitus with complications;
16. History of thrombocytopenia or other coagulation disorders, which may cause intramuscular injection contraindications;
17. Abnormal and uncontrolled blood pressure during physical examination before vaccination (for subjects aged 40-59: systolic pressure ≥ 140 mmHg and/or diastolic pressure ≥ 90 mmHg; for subjects aged ≥60, systolic pressure ≥ 150 mmHg and/or diastolic pressure ≥ 100 mmHg);
18. History of drug abuse (narcotic drugs, psychotropic drugs);
19. Patients with previous or current malignant tumors (except papillary thyroid cancer);
20. Receipt of investigational or unapproved products (drugs or vaccines) within 6 months before vaccination; or planned participation in another clinical study during the study period;
21. Any condition that, in the opinion the investigator, makes subjects ineligible for the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2024-12-09 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
The geometric mean concentration (GMC) of anti-gE antibodies one month after full vaccination. | At Month 0 and Month 3.
  Anti-gE antibody concentrations, were determined by ELISA, expressed as Geometric Mean Concentrations (GMCs), in milli international units per milliliter.

SECONDARY OUTCOMES:
The seroconversion rate of anti-gE antibodies one month after full vaccination. | At Month 3.
  Vaccine response was defined as: For initially seronegative subjects, antibody concentration at post-vaccination ≥ 4 fold the cut-off for Anti-gE; For initially seropositive subjects, antibody concentration at post-vaccination ≥ 4 fold the pre-vaccination antibody concentration.
The incidence, severity, and vaccine-related association of solicited local adverse events (AEs) within 7 days after each dose of vaccination. | During the 7 days (Days 0-6) after each vaccine dose.
  This typically refers to the documentation and assessment of local adverse events (such as pain and swelling at the injection site) that occur within 7 days after vaccination in clinical studies or vaccination programs. This includes the frequency of occurrence, severity (usually categorized as mild, moderate, and severe), and the investigator's assessment of the association between these events and vaccination.
The incidence, severity, and relevance to vaccination of solicited general adverse events (AEs) within 7 days after each dose of vaccination. | During the 7 days (Days 0-6) after each vaccine dose.
  This typically refers to the documentation and assessment of general adverse events that occur within the 7-day observation period after each vaccination dose, including the frequency of occurrence, severity (such as mild, moderate, and severe), and the investigator's assessment of the association between these events and the vaccination.
The incidence, severity, and relevance to vaccination of unsolicited adverse events (AEs) within 30 days after each vaccine dose. | During 30 days (Days 0-29) after each vaccination.
  This typically refers to the documentation and assessment of unexpected adverse events that occur within the 30-day observation period after each vaccine dose, including the frequency of occurrence, severity (such as mild, moderate, and severe), and the investigator's assessment of the association between these events and vaccination.
The incidence of serious adverse events (SAEs) from the first dose of vaccination to one month after the final dose. | From first vaccination up to 30 days post last vaccination (Month 0-Month 3).
  Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
The incidence of potential immune-mediated diseases (pIMDs) from the first dose of vaccination to one month after the final dose. | From first vaccination up to 30 days post last vaccination (Month 0-Month 3).
  Potential immune-mediated diseases (pIMDs) are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.

CONTACTS AND LOCATIONS:
Overall Officials: Yanxia Wang, Master, Principal Investigator — Henan Center for Disease Control and Prevention
Locations (1):
- Henan Center for Diseases Control and Prevention, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No